CLINICAL TRIAL: NCT01930422
Title: Effect of Transcranial Direct Current Stimulation (tDCS) on Tobacco Consumption.
Acronym: TABELEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12 392 02; AOL 2012 (Other: Toulouse University Hospital)
Record Dates: First submitted 2013-06-20; First posted 2013-08-29 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Tobacco Use Disorder
Keywords: Direct transcranial electrical stimulation (tDCS); Sham procedure; Tobacco consumption; Craving
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real tDCS (Experimental): Direct transcranial electrical stimulation (tDCS procedure)
  Interventions: Device: tDCS procedure
- Placebo tDCS (Sham Comparator): Sham procedure
  Interventions: Device: Sham procedure

INTERVENTIONS:
Device: tDCS procedure — The tDCS is a non-invasive neuromodulation method. A stimulator delivers a constant current of low intensity (1-2 mA) applied to the average of two bipolar electrodes placed on the scalp for 20 minutes. This constant current generates a static electric field that selectively modulates the activity of cortical neurones. A tingling sensation under the electrodes appears at the beginning and at the end of stimulation but it is transient and disappears quickly in 30 or 60 seconds.
  Arms: Real tDCS
Device: Sham procedure — The tDCS placebo differs from the real tDCS by the interruption of stimulation after 30 to 60 seconds and reactivation of this stimulation 30 to 60 seconds before the end of the session, which lasted 20 minutes. The tingling felt at the beginning and the end of the session will be the same as those experienced with real stimulation. The electrodes establishment does not differ with respect to tDCS.
  Arms: Placebo tDCS

SUMMARY:
The primary purpose of the protocol is to evaluate the effect of repeated application for 5 consecutive days of a real tDCS compared to the application of a placebo tDCS (sham procedure) on the evolution of tobacco consumption in the short term between Day 1 and Day 5.

The study hypothesis is that a repeated application for 5 consecutive days of a real tDCS on the left dorsolateral prefrontal cortex region will reduce the craving induced causing a decreased of daily tobacco consumption between Day 1 and Day 5 which can persist at the final visit between Day 15 and Day 20.

DETAILED DESCRIPTION:
Smoking is a major public health problem and it is the leading cause of preventable death in the world. Care should include education, psychotherapy and treatments, but despite these therapeutics, the smoking cessation process is often characterized by relapses. The main risk factor for relapse is craving. Neurophysiological studies have provided evidence in the understanding of craving. This craving involves surface structures including the dorsolateral prefrontal cortex, accessible by neurostimulation. Repetitive neurostimulation applies on this structures involved in craving could therefore modulate it. Two non-invasive stimulation techniques exist: repetitive transcranial magnetic stimulation (rTMS) and transcranial direct current stimulation (tDCS). The choice of tDCS is based on its ease of use, excellent tolerance, its better quality of placebo and low cost.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 60 years old
* Smoking ≥ 5 years
* Smoking ≥ 15 manufactured cigarettes per day or ≥ 10 rolled cigarettes per day
* Fagerström test ≥ 5
* Smokers who have at least an attempt to stop of minimum 7 days
* Written informed consent signed by the patient
* Affiliated to medical insurance

Exclusion Criteria:

* Co-addiction (cannabis, alcohol, other drugs)
* HAD test: D ≥ 8; A + D ≥ 19
* Treatment by nicotine replacement therapy, bupropion or varenicline within 30 days prior inclusion
* Neuropsychiatric disease, considered serious by the investigator
* Psychotropic treatment (antidepressant, anxiolytic, antipsychotic)
* Skin scalp dermatosis
* Pregnancy or breastfeeding. Positive pregnancy test.
* Patient under guardianship, trusteeship or judicial protection
* Patient in inclusion period for another clinical research protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2013-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Relative change of individual salivary cotinine. | Outcome measure is assessed at Day1 and Day5

SECONDARY OUTCOMES:
Relative change of individual salivary cotinine | Outcome measure is assessed at Day5 and between Day15 and Day20.
Exhaled carbon monoxide. | Outcome measure is assessed at day 0, day 1, day 2, day 3, day 4, day 5 and between day 15 and day 20.
Number of cigarettes smoked per day | Outcome measure is assessed at day 0, day1, day2, day3, day4, day5 and between day 15 and 20
Technical feasibility of outpatient | Outcome measure is assessed between day 15 and 20.
  The feasibility is assessed by the number of smokers following the entire protocol.
Measurement of craving | Outcome measure is assessed at Day1, day2, day3, day4, day5 and betwenn day 15 to day 20.
  Measurement of craving from Day1 to Day5 and at the final visits assessed by a VAS: visual analogue scale from 0 (no urge to smoke at all) to 10 (intense desire compelling smoking) and the questionnaire called the 12-item French Tobacco Craving Questionnaire (FCTQ-12).

CONTACTS AND LOCATIONS:
Overall Officials: Rose-Marie ROUQUET, MD, Principal Investigator
Locations (1):
- University Hospital, Toulouse, Toulouse, Midi-Pyrénées, France

REFERENCES:
- [Background] Organisation Mondiale de la Santé. Rapport de l'OMS sur l'épidémie mondiale de tabagisme 2011, résumé d'orientation. OMS 2011
- [Background] Rapport OMS Mpower 2008.
- [Background] Observatoire français des drogues et des toxicomanies. Les niveaux d'usage des drogues en France en 2010. OFDT Tendances, n°76, juin 2011
- [Background] Le Faou AL, Scemama O. [Epidemiology of tobacco smoking]. Rev Mal Respir. 2005 Dec;22(6 Pt 2):8S27-32. French. PMID 16340832
- [Background] Hill C, Jougla E, Beck F. Le point sur l'épidémie de cancer du poumon dû au tabagisme. BEH mai 2010; 19-20: 210-213
- [Background] Fuxe, K., Anderson, K., Eneroth, P., 1987. Effects of nicotine and exposure to cigarette smoke on discrete dopamine and noradrenaline nerve terminal systems of the telcephalon and diencephalon of the rat: relationship to reward mechanisms and distribution of nicotine binding sites in brain. In: Martin, W.R., Van Loon, G.R., Iwamoto, E.T., et al. (Eds.), Tobacco Smoking and Nicotine: A Neurobiological Approach. Plenum, New York, pp. 225-262.
- [Background] Pert, A., Clarke, P.B.S., 1987. Nicotine modulation of dopaminergic transmission: functional implications. In: Martin, W.R., Van Loon, G.R., Iwamoto, E.T., et al. (Eds.), Tobacco, Smoking and Nicotine: A Neurobiological Approach. Plenum, New York, pp.169-189.
- [Background] United States Department of Health and Human Services, 1988. The Health Consequences of Smoking: Nicotine Addiction. US Government Printing Office, Washington, DC DHHS Publication No.CDC-88-8406.
- [Background] Clarke, P., 1990. Mesolimbic dopaminergic activation: the key to nicotine reinforcement. In: Bock, G., Marsh, J. (Eds.), The Biology of Nicotine Dependence. Wiley, New York, pp. 153-168.
- [Background] Pich EM, Pagliusi SR, Tessari M, Talabot-Ayer D, Hooft van Huijsduijnen R, Chiamulera C. Common neural substrates for the addictive properties of nicotine and cocaine. Science. 1997 Jan 3;275(5296):83-6. doi: 10.1126/science.275.5296.83. PMID 8974398
- [Background] Wise RA, Bozarth MA. A psychomotor stimulant theory of addiction. Psychol Rev. 1987 Oct;94(4):469-92. No abstract available. PMID 3317472
- [Background] Collins AC, Marks MJ. Progress towards the development of animal models of smoking-related behaviors. J Addict Dis. 1991;10(1-2):109-26. doi: 10.1300/J069v10n01_08. PMID 2065112
- [Background] Pomerleau OF. Individual differences in sensitivity to nicotine: implications for genetic research on nicotine dependence. Behav Genet. 1995 Mar;25(2):161-77. doi: 10.1007/BF02196925. PMID 7733857
- [Background] Robinson TE, Berridge KC. The neural basis of drug craving: an incentive-sensitization theory of addiction. Brain Res Brain Res Rev. 1993 Sep-Dec;18(3):247-91. doi: 10.1016/0165-0173(93)90013-p. PMID 8401595
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Background] Pickens RW, Johanson CE. Craving: consensus of status and agenda for future research. Drug Alcohol Depend. 1992 Jun;30(2):127-31. doi: 10.1016/0376-8716(92)90017-7. PMID 1633752
- [Background] Marlatt, G.A., Gordon, J.R. (Eds.), 1985. Relapse Prevention. Guilford, New York
- [Background] Killen JD, Fortmann SP. Craving is associated with smoking relapse: findings from three prospective studies. Exp Clin Psychopharmacol. 1997 May;5(2):137-42. doi: 10.1037//1064-1297.5.2.137. PMID 9234050
- [Background] Shiffman S, Engberg JB, Paty JA, Perz WG, Gnys M, Kassel JD, Hickcox M. A day at a time: predicting smoking lapse from daily urge. J Abnorm Psychol. 1997 Feb;106(1):104-16. doi: 10.1037//0021-843x.106.1.104. PMID 9103722
- [Background] Abrams DB, Monti PM, Pinto RP, Elder JP, Brown RA, Jacobus SI. Psychosocial stress and coping in smokers who relapse or quit. Health Psychol. 1987;6(4):289-303. doi: 10.1037//0278-6133.6.4.289. PMID 3301320
- [Background] Niaura R, Abrams DB, Pedraza M, Monti PM, Rohsenow DJ. Smokers' reactions to interpersonal interaction and presentation of smoking cues. Addict Behav. 1992 Nov-Dec;17(6):557-66. doi: 10.1016/0306-4603(92)90065-4. PMID 1488936
- [Background] Shiffman S, Paty JA, Gnys M, Kassel JA, Hickcox M. First lapses to smoking: within-subjects analysis of real-time reports. J Consult Clin Psychol. 1996 Apr;64(2):366-79. doi: 10.1037//0022-006x.64.2.366. PMID 8871421
- [Background] Brody AL, Mandelkern MA, London ED, Childress AR, Lee GS, Bota RG, Ho ML, Saxena S, Baxter LR Jr, Madsen D, Jarvik ME. Brain metabolic changes during cigarette craving. Arch Gen Psychiatry. 2002 Dec;59(12):1162-72. doi: 10.1001/archpsyc.59.12.1162. PMID 12470133
- [Background] McClernon FJ, Hiott FB, Huettel SA, Rose JE. Abstinence-induced changes in self-report craving correlate with event-related FMRI responses to smoking cues. Neuropsychopharmacology. 2005 Oct;30(10):1940-7. doi: 10.1038/sj.npp.1300780. PMID 15920499
- [Background] Wilson SJ, Sayette MA, Delgado MR, Fiez JA. Instructed smoking expectancy modulates cue-elicited neural activity: a preliminary study. Nicotine Tob Res. 2005 Aug;7(4):637-45. doi: 10.1080/14622200500185520. PMID 16085533
- [Background] Smolka MN, Buhler M, Klein S, Zimmermann U, Mann K, Heinz A, Braus DF. Severity of nicotine dependence modulates cue-induced brain activity in regions involved in motor preparation and imagery. Psychopharmacology (Berl). 2006 Mar;184(3-4):577-88. doi: 10.1007/s00213-005-0080-x. Epub 2005 Aug 13. PMID 16133128
- [Background] Brody AL, Mandelkern MA, Olmstead RE, Jou J, Tiongson E, Allen V, Scheibal D, London ED, Monterosso JR, Tiffany ST, Korb A, Gan JJ, Cohen MS. Neural substrates of resisting craving during cigarette cue exposure. Biol Psychiatry. 2007 Sep 15;62(6):642-51. doi: 10.1016/j.biopsych.2006.10.026. Epub 2007 Jan 9. PMID 17217932
- [Background] Lee JH, Lim Y, Wiederhold BK, Graham SJ. A functional magnetic resonance imaging (FMRI) study of cue-induced smoking craving in virtual environments. Appl Psychophysiol Biofeedback. 2005 Sep;30(3):195-204. doi: 10.1007/s10484-005-6377-z. PMID 16167185
- [Background] Due DL, Huettel SA, Hall WG, Rubin DC. Activation in mesolimbic and visuospatial neural circuits elicited by smoking cues: evidence from functional magnetic resonance imaging. Am J Psychiatry. 2002 Jun;159(6):954-60. doi: 10.1176/appi.ajp.159.6.954. PMID 12042183
- [Background] Ferguson SG, Shiffman S. The relevance and treatment of cue-induced cravings in tobacco dependence. J Subst Abuse Treat. 2009 Apr;36(3):235-43. doi: 10.1016/j.jsat.2008.06.005. Epub 2008 Aug 20. PMID 18715743
- [Background] Tiffany ST, Cox LS, Elash CA. Effects of transdermal nicotine patches on abstinence-induced and cue-elicited craving in cigarette smokers. J Consult Clin Psychol. 2000 Apr;68(2):233-40. doi: 10.1037//0022-006x.68.2.233. PMID 10780123
- [Background] Singleton EG, Anderson LM, Heishman SJ. Reliability and validity of the Tobacco Craving Questionnaire and validation of a craving-induction procedure using multiple measures of craving and mood. Addiction. 2003 Nov;98(11):1537-46. doi: 10.1046/j.1360-0443.2003.00449.x. PMID 14616180
- [Background] Heishman SJ, Singleton EG, Moolchan ET. Tobacco Craving Questionnaire: reliability and validity of a new multifactorial instrument. Nicotine Tob Res. 2003 Oct;5(5):645-54. doi: 10.1080/1462220031000158681. PMID 14577981
- [Background] Berlin I, Vorspan F, Singleton EG, Warot D, Notides C, Heishman SJ. Reliability and validity of the French version of the tobacco craving questionnaire. Eur Addict Res. 2005;11(2):62-8. doi: 10.1159/000083034. PMID 15785066
- [Background] Heishman SJ, Singleton EG, Pickworth WB. Reliability and validity of a Short Form of the Tobacco Craving Questionnaire. Nicotine Tob Res. 2008 Apr;10(4):643-51. doi: 10.1080/14622200801908174. PMID 18418787
- [Background] Berlin I, Singleton EG, Heishman SJ. Validity of the 12-item French version of the Tobacco Craving Questionnaire in treatment-seeking smokers. Nicotine Tob Res. 2010 May;12(5):500-7. doi: 10.1093/ntr/ntq039. Epub 2010 Mar 24. PMID 20335281
- [Background] Koob GF, Sanna PP, Bloom FE. Neuroscience of addiction. Neuron. 1998 Sep;21(3):467-76. doi: 10.1016/s0896-6273(00)80557-7. No abstract available. PMID 9768834
- [Background] Afssaps 2003 (RBPC) : stratégies thérapeutiques médicamenteuses et non médicamenteuses de l'aide à l'arrêt du tabac
- [Background] Stead LF, Perera R, Bullen C, Mant D, Lancaster T. Nicotine replacement therapy for smoking cessation. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD000146. doi: 10.1002/14651858.CD000146.pub3. PMID 18253970
- [Background] Woolacott NF, Jones L, Forbes CA, Mather LC, Sowden AJ, Song FJ, Raftery JP, Aveyard PN, Hyde CJ, Barton PM. The clinical effectiveness and cost-effectiveness of bupropion and nicotine replacement therapy for smoking cessation: a systematic review and economic evaluation. Health Technol Assess. 2002;6(16):1-245. doi: 10.3310/hta6160. No abstract available. PMID 12269277
- [Background] Silagy C, Lancaster T, Stead L, Mant D, Fowler G. Nicotine replacement therapy for smoking cessation. Cochrane Database Syst Rev. 2004;(3):CD000146. doi: 10.1002/14651858.CD000146.pub2. PMID 15266423
- [Background] Hughes JR, Stead LF, Lancaster T. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2007 Jan 24;(1):CD000031. doi: 10.1002/14651858.CD000031.pub3. PMID 17253443
- [Background] Moore TJ, Furberg CD, Glenmullen J, Maltsberger JT, Singh S. Suicidal behavior and depression in smoking cessation treatments. PLoS One. 2011;6(11):e27016. doi: 10.1371/journal.pone.0027016. Epub 2011 Nov 2. PMID 22073240
- [Background] Cahill K, Stead LF, Lancaster T. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2007 Jan 24;(1):CD006103. doi: 10.1002/14651858.CD006103.pub2. PMID 17253581
- [Background] Afssaps - Plan de gestion de risque de la spécialité pharmaceutique CHAMPIX ® Fev 2008
- [Background] Gourlay SG, Stead LF, Benowitz NL. Clonidine for smoking cessation. Cochrane Database Syst Rev. 2004;2004(3):CD000058. doi: 10.1002/14651858.CD000058.pub2. PMID 15266422
- [Background] Public Health Service. Treating tobacco use and dependence. Clinical practice guideline. Washington (DC):US Department of Health and Human Services; 2000.
- [Background] Raupach T, Hoogsteder PH, Onno van Schayck CP. Nicotine vaccines to assist with smoking cessation: current status of research. Drugs. 2012 Mar 5;72(4):e1-16. doi: 10.2165/11599900-000000000-00000. PMID 22356293
- [Background] Cottraux J. Les thérapies comportementales et cognitives, 4ème édition Historique Masson 2004; 2: 20-32
- [Background] Cottraux J. Les thérapies comportementales et cognitives, 4ème édition Des théories de l'apprentissage aux théories cognitives Masson 2004; 3: 35-66
- [Background] Le Foll B, Aubin HJ, Lagrue G. [Behavioral and cognitive therapy to break the smoking habit. Review of the literature]. Ann Med Interne (Paris). 2002 May;153(3 Suppl):1S32-40. French. PMID 12218881
- [Background] Avis de la HAS, Haute Autorité de Santé Stratégies thérapeutiques d'aide au sevrage tabagique, efficacité, efficience et prise en charge financière. HAS, octobre 2006
- [Background] Agence Française de Sécurité Sanitaire des Produits de Santé Les stratégies thérapeutiques médicamenteuses et non médicamenteuses de l'aide à l'arrêt du tabac. Argumentaire, Recommandations de bonne pratique. AFSSAPS, mai 2003
- [Background] Lang N, Hasan A, Sueske E, Paulus W, Nitsche MA. Cortical hypoexcitability in chronic smokers? A transcranial magnetic stimulation study. Neuropsychopharmacology. 2008 Sep;33(10):2517-23. doi: 10.1038/sj.npp.1301645. Epub 2007 Dec 5. PMID 18059439
- [Background] Brunelin J, Poulet E, Boeuve C, Zeroug-vial H, d'Amato T, Saoud M. [Efficacy of repetitive transcranial magnetic stimulation (rTMS) in major depression: a review]. Encephale. 2007 Mar-Apr;33(2):126-34. doi: 10.1016/s0013-7006(07)91542-0. French. PMID 17675907
- [Background] Meng Z, Liu S, Zheng Y, Phillips JS. Repetitive transcranial magnetic stimulation for tinnitus. Cochrane Database Syst Rev. 2011 Oct 5;(10):CD007946. doi: 10.1002/14651858.CD007946.pub2. PMID 21975776
- [Background] Barr MS, Fitzgerald PB, Farzan F, George TP, Daskalakis ZJ. Transcranial magnetic stimulation to understand the pathophysiology and treatment of substance use disorders. Curr Drug Abuse Rev. 2008 Nov;1(3):328-39. doi: 10.2174/1874473710801030328. PMID 19630729
- [Background] Hoppner J, Broese T, Wendler L, Berger C, Thome J. Repetitive transcranial magnetic stimulation (rTMS) for treatment of alcohol dependence. World J Biol Psychiatry. 2011 Sep;12 Suppl 1:57-62. doi: 10.3109/15622975.2011.598383. PMID 21905997
- [Background] Barth KS, Rydin-Gray S, Kose S, Borckardt JJ, O'Neil PM, Shaw D, Madan A, Budak A, George MS. Food cravings and the effects of left prefrontal repetitive transcranial magnetic stimulation using an improved sham condition. Front Psychiatry. 2011 Mar 14;2:9. doi: 10.3389/fpsyt.2011.00009. eCollection 2011. PMID 21556279
- [Background] Johann M, Wiegand R, Kharraz A, Bobbe G, Sommer G, Hajak G, Wodarz N, Eichhammer P. [Repetitiv Transcranial Magnetic Stimulation in Nicotine Dependence]. Psychiatr Prax. 2003 May;30(Suppl 2):129-131. doi: 10.1055/s-2003-39733. German. PMID 13130356
- [Background] Eichhammer P, Johann M, Kharraz A, Binder H, Pittrow D, Wodarz N, Hajak G. High-frequency repetitive transcranial magnetic stimulation decreases cigarette smoking. J Clin Psychiatry. 2003 Aug;64(8):951-3. doi: 10.4088/jcp.v64n0815. PMID 12927012
- [Background] Amiaz R, Levy D, Vainiger D, Grunhaus L, Zangen A. Repeated high-frequency transcranial magnetic stimulation over the dorsolateral prefrontal cortex reduces cigarette craving and consumption. Addiction. 2009 Apr;104(4):653-60. doi: 10.1111/j.1360-0443.2008.02448.x. Epub 2009 Jan 12. PMID 19183128
- [Background] Rose JE, McClernon FJ, Froeliger B, Behm FM, Preud'homme X, Krystal AD. Repetitive transcranial magnetic stimulation of the superior frontal gyrus modulates craving for cigarettes. Biol Psychiatry. 2011 Oct 15;70(8):794-799. doi: 10.1016/j.biopsych.2011.05.031. Epub 2011 Jul 18. PMID 21762878
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] Nitsche MA, Cohen LG, Wassermann EM, Priori A, Lang N, Antal A, Paulus W, Hummel F, Boggio PS, Fregni F, Pascual-Leone A. Transcranial direct current stimulation: State of the art 2008. Brain Stimul. 2008 Jul;1(3):206-23. doi: 10.1016/j.brs.2008.06.004. Epub 2008 Jul 1. PMID 20633386
- [Background] Gartside IB. Mechanisms of sustained increases of firing rate of neurones in the rat cerebral cortex after polarization: role of protein synthesis. Nature. 1968 Oct 26;220(5165):383-4. doi: 10.1038/220383a0. No abstract available. PMID 4300961
- [Background] Hattori Y, Moriwaki A, Hori Y. Biphasic effects of polarizing current on adenosine-sensitive generation of cyclic AMP in rat cerebral cortex. Neurosci Lett. 1990 Aug 24;116(3):320-4. doi: 10.1016/0304-3940(90)90094-p. PMID 2173816
- [Background] Islam N, Aftabuddin M, Moriwaki A, Hattori Y, Hori Y. Increase in the calcium level following anodal polarization in the rat brain. Brain Res. 1995 Jul 3;684(2):206-8. doi: 10.1016/0006-8993(95)00434-r. PMID 7583224
- [Background] Gandiga PC, Hummel FC, Cohen LG. Transcranial DC stimulation (tDCS): a tool for double-blind sham-controlled clinical studies in brain stimulation. Clin Neurophysiol. 2006 Apr;117(4):845-50. doi: 10.1016/j.clinph.2005.12.003. Epub 2006 Jan 19. PMID 16427357
- [Background] Bikson M, Datta A, Elwassif M. Establishing safety limits for transcranial direct current stimulation. Clin Neurophysiol. 2009 Jun;120(6):1033-4. doi: 10.1016/j.clinph.2009.03.018. Epub 2009 Apr 24. No abstract available. PMID 19394269
- [Background] Poreisz C, Boros K, Antal A, Paulus W. Safety aspects of transcranial direct current stimulation concerning healthy subjects and patients. Brain Res Bull. 2007 May 30;72(4-6):208-14. doi: 10.1016/j.brainresbull.2007.01.004. Epub 2007 Jan 24. PMID 17452283
- [Background] Fregni F, Liguori P, Fecteau S, Nitsche MA, Pascual-Leone A, Boggio PS. Cortical stimulation of the prefrontal cortex with transcranial direct current stimulation reduces cue-provoked smoking craving: a randomized, sham-controlled study. J Clin Psychiatry. 2008 Jan;69(1):32-40. doi: 10.4088/jcp.v69n0105. PMID 18312035
- [Background] Boggio PS, Liguori P, Sultani N, Rezende L, Fecteau S, Fregni F. Cumulative priming effects of cortical stimulation on smoking cue-induced craving. Neurosci Lett. 2009 Sep 29;463(1):82-6. doi: 10.1016/j.neulet.2009.07.041. Epub 2009 Jul 18. PMID 19619607
- [Background] Boggio PS, Zaghi S, Villani AB, Fecteau S, Pascual-Leone A, Fregni F. Modulation of risk-taking in marijuana users by transcranial direct current stimulation (tDCS) of the dorsolateral prefrontal cortex (DLPFC). Drug Alcohol Depend. 2010 Dec 1;112(3):220-5. doi: 10.1016/j.drugalcdep.2010.06.019. Epub 2010 Aug 21. PMID 20729009
- [Background] Boggio PS, Sultani N, Fecteau S, Merabet L, Mecca T, Pascual-Leone A, Basaglia A, Fregni F. Prefrontal cortex modulation using transcranial DC stimulation reduces alcohol craving: a double-blind, sham-controlled study. Drug Alcohol Depend. 2008 Jan 1;92(1-3):55-60. doi: 10.1016/j.drugalcdep.2007.06.011. Epub 2007 Jul 19. PMID 17640830
- [Background] Fu M, Fernandez E, Martinez-Sanchez JM, Pascual JA, Schiaffino A, Agudo A, Ariza C, Borras JM, Samet JM; DCOT Study investigators. Salivary cotinine concentrations in daily smokers in Barcelona, Spain: a cross-sectional study. BMC Public Health. 2009 Sep 3;9:320. doi: 10.1186/1471-2458-9-320. PMID 19728886
- [Background] Fu M, Martinez-Sanchez JM, Agudo A, Pascual JA, Ariza C, Moncada A, Fernandez E; DCOT Study Investigators. Nicotine depedence and salivary cotinine concentration in daily smokers. Eur J Cancer Prev. 2012 Jan;21(1):96-102. doi: 10.1097/CEJ.0b013e32834a7e59. PMID 22129659